CLINICAL TRIAL: NCT05331807
Title: The Effects of Combined Omega-3 and Vitamin D Supplementation on Nutritional Status, Quality of Life and Inflammatory Markers Among the Breast Cancer Women in Gaza Strip
Brief Title: Omega-3 and Vitamin D Supplementation in Breast Cancer Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Leng Huat Foo, Associate Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21090645
Record Dates: First submitted 2022-03-18; First posted 2022-04-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: An open-label randomized clinical trial of breast cancer women that are undergoing chemotherapy treatment for total duration of 2 months (approximately 9 weeks in total), in which participants will be randomly selected and included in either one of these four (4) experimental groups (arms).
Masking Description: All eligible participants will be randomly selected and included in either one of these four (4) experimental groups (arms).The participants for each experimental will matched and stratified based on age group (± 5 years), menopausal status and BMI status (± 2 kg/m2). Each participant will be randomly allocated into four groups, based on their age, menopausal status and BMI status to ensure the standardization of general characteristics of study participants included in the study as a baseline data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (A) (Experimental): Participants will be received daily omega-3 fatty acid (two capsules of 1000mg fish oil daily). Each soft gel capsule contains 300 mg of omega-3 fatty acids in the bioactive triglyceride (TG) and 180mg EPA and 120 mg DHA. (Omega3 complex, Jamieson Laboratories, Canada)
  Interventions: Dietary Supplement: Omega-3 FA
- Group (B) (Experimental): Participants will be received only vitamin D (one capsule of 50,000IU weekly). Each film coated tablet of vitamin D contains 50,000 IU Vitamin D3 (Cholecalciferol). (J-Dee, Jerusalem Pharmaceutical Company, West bank, Palestine).
  Interventions: Dietary Supplement: Vitamin D
- Group (C) (Experimental): Participants will be received both omega-3 fatty acids capsules and vitamin D3 capsule. (one capsule of D3 50,000 IU weekly + two omega-3 fatty acids capsules daily (each capsule contains 300 mg of omega-3 fatty acids)
  Interventions: Combination Product: Combined Omega-3 and Vitamin D Supplementation
- Group (D) (No Intervention): Participants will not be received any supplements and just receive oncology treatment as an usual oncology patient.

INTERVENTIONS:
Dietary Supplement: Omega-3 FA — Two capsules of 1000mg fish oil daily (Each soft gel capsule contains 180mg EPA and 120 mg DHA)
  Arms: Group (A)
Dietary Supplement: Vitamin D — one capsule of vitamin D3 weekly (one D3 capsule contains 50,000 IU)
  Arms: Group (B)
Combination Product: Combined Omega-3 and Vitamin D Supplementation — Two capsules of 1000mg fish oil daily (Each soft gel capsule contains 180mg EPA and 120 mg DHA) and one capsule of vitamin D3 weekly (one D3 capsule contains 50,000 IU)
  Arms: Group (C)

SUMMARY:
Breast cancer (BC) is the most common malignant disease, which is fifth leading cause of cancer mortality worldwide. Poor nutritional status is one of the common physical symptoms found among cancer patients, in which it is caused by both cancer disease state and its oncology treatment regimens used. Cancer patients develop a tumor-associated malnutrition characterized by an insufficient supply of macro- and micronutrients and systemic chemotherapy treatment that could significantly affecting the nutritional status of these patients by its side effects associated with chemotherapy that may lead to many medical complications that often requires hospitalization and death. An adequate nutritional intervention can have a beneficial impact on the disease condition and also the progress of the disease, as an integral part of adjuvant therapy on cancer care. Numerous studies had shown that the use of EPA and DHA are safe (absence of cardiotoxic effects) and effective in reducing the common chemotherapy-related side effects, such as bone density loss, peripheral neuropathy and weight gain. The question remains arises to whether administration of both vitamin D and omega-3 fatty acids supplementations could be used as important nutritional strategy during the active oncology treatment in breast cancer patients. In Palestine, nutritional intervention strategies are poorly evaluated in the oncology setting especially among patients undergoing chemotherapy. Suitable and proper nutritional interventions among breast cancer patients during active oncology treatments could help to improve nutritional status, decrease mortality and improve quality of life among these subjects. Hence, the present study is formulated to assess the effect of combined omega-3 fatty acid and vitamin D supplementation on the nutritional status, quality of life and blood inflammatory markers among breast cancer women undergoing chemotherapy treatment in the Gaza Strip, Palestine.

DETAILED DESCRIPTION:
An adequate nutritional intervention can have a beneficial impacts on the disease condition and also the progress of the disease, as an integral part of adjuvant therapy on cancer care. Numerous clinical and epidemiological studies had found that vitamin D deficiency is common nutritional disorder in BC patients and that significantly associated with a negative prognostic factor, in which some have reported a positive effect of combining vitamin D or its analogues as an adjuvant therapy, together with a variety of chemotherapeutic factors used during oncology treatments. Moreover, combination of vitamin D and omega-3 fatty acids may provide a new complementary treatment by decreasing inflammatory biomarkers and resistance to cancer treatment in patients with BC. The question remains whether vitamin D and omega-3 fatty acids co-supplementation would actually be useful after diagnosis of BC. So, the aim of this study is to investigate the effects of vitamin D and omega-3 fatty acids co-supplementation on inflammatory biomarkers, and nutritional status in patients with BC.

ELIGIBILITY:
Inclusion Criteria:

* Females who have been newly diagnosed with the breast cancer of stage I, II and III
* Patients with following clinical diagnosis of breast cancer such as lymph node positive +ve, hormonal receptor negative -ve and human epidermal growth factor receptor 2 (HER2) negative -ve
* Patient will receive her first chemotherapy treatment with Adriamycin + Cytoxan (AC) for a total of four cycle (each cycle will be carried-out every 3 weeks (21 days)

Exclusion Criteria:

* Participants who had already undertaken her chemotherapy previously, and/or other oncology treatments such as hormonal or radiation oncology therapy
* Patients with recurrent breast cancer, patients with other chronic disease conditions such as renal disease and under dialysis, HIV, malabsorption disorder diseases, autoimmune diseases, diabetes, hypertension, hepatic, parathyroid, and gastrointestinal disorders.
* Patients who have reported any allergy condition to fish and/or fish products
* Pregnant women

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breast cancer patients
Enrollment: 88 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change of Nutritional status, as assessed by Body Mass Index | Change from Baseline BMI at 2 months
  Body weight in kilograms and height in meters will be combined to report BMI in kg/m^2
Change of body weight | Change from Baseline Weight in kg at 2 months
  Body weight will be measured in kilograms
Change of Muscle Mass Status | Change from Baseline calf circumference in cm at 2 months
  Muscle mass status will be assessed by calf circumference levels in cm. Higher values of calf circumference is indicative of greater lean mass.
Change of Nutritional Status Condition, as assessed by the Patient-Generated Subjective Global Assessment PG-SGA | Change from Baseline Nutritional Status Condition in category of well-nourished, moderately malnourished or severely malnourished at 2 months
  The PG-SGA will be based four components such as questions related to body weight status (scored 0-5), food intake (score 0-4); symptoms affecting oral food intake (scored 0-23), and lastly questions on daily activities and function, in which the degree of malnutrition of patients will be classified as (A) well-nourished; (B) moderately malnourished; or (C) severely malnourished.
Change of Total Scale and Single-item measures Scores derived from the Quality of life questionnaire (QLQ C-30) assessment | Change from Baseline total scales and single-item measures scores (0 to 100 scores) at 2 months
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) assessment of 30 questions to measure cancer patients' physical, psychological and social functions. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Change of Blood inflammatory markers of blood TNF-α levels | Change from baseline TNF-α levels in pg/mL at 2 months
  Blood concentration of TNF-α levels will be measured in unit pg/mL.
Change of Blood inflammatory markers of blood CRP levels | Change from baseline CRP levels in nmol/L at 2 months
  Blood concentration of CRP levels will be measured in nmol/L
Change of Nutritional Status Assessed by body weight levels | Change from baseline weight in kg at 2 months
  Body weight will be measured in kilograms

SECONDARY OUTCOMES:
Change of Dietary Energy Intakes | Change from Baseline dietary energy intakes in kcal at 2 months
  Habitual dietary nutrients intake will be assessed by mean energy intakes in kcal
Change of Dietary Fat Intakes | Change from Baseline dietary fat intakes in grams at 2 months
  Habitual dietary nutrients intake will be assessed by mean fat intakes in grams
Change of Dietary Protein Intakes | Change from Baseline dietary Protein intakes in grams at 2 months
  Habitual dietary protein intakes will be assessed by mean protein intakes in grams
Change of Dietary Vitamin D intakes | Change from Baseline Dietary Vitamin D Intakes in microgram at 2 months
  Habitual dietary nutrients intake will be assessed by mean vitamin D intakes in micrograms
Lifestyle physical activity status | Change from Baseline Physical Activity Status (inactive, minimally active or active physical activity status) at 2 months
  A short form of the international physical activity questionnaire (IPAQ) will be used to assess the physical activity levels of the study participants, in which three different category groups of inactive, minimally active and active will be categorised.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkish-Palestinian Friendship Hospital, Al-Zahra', Gaza Strip, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almassri HF, Abdul Kadir A, Srour M, Foo LH. The Effects of Omega-3 Fatty Acids and Vitamin D Supplementation on the Nutritional Status of Women with Breast Cancer in Palestine: An Open-Label Randomized Controlled Trial. Nutrients. 2024 Nov 20;16(22):3960. doi: 10.3390/nu16223960. PMID 39599746
- [Derived] Almassri HF, Abdul Kadir A, Srour M, Foo LH. The effects of Omega-3 fatty acids and vitamin D supplementation on the quality of life and blood inflammation markers in newly diagnosed breast cancer women: An open-labelled randomised controlled trial. Clin Nutr ESPEN. 2025 Feb;65:64-75. doi: 10.1016/j.clnesp.2024.11.014. Epub 2024 Nov 20. PMID 39577691